CLINICAL TRIAL: NCT06356025
Title: Botulinum Toxin Injection in the Upper Esophageal Sphincter for Retrograde-cricopharyngeus Dysfunction: a Prospective, Double Blind, Placebo-controlled Trial
Brief Title: Botulinum Toxin Injection in the UES for R-CPD
Acronym: BOTUS R-CPD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Delta (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 52082; 2024-512546-42 (EudraCT Number)
Record Dates: First submitted 2024-03-20; First posted 2024-04-10 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Retrograde Cricopharyngeus Dysfunction
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin injection (Experimental)
  Interventions: Drug: botulinum toxin type A
- Placebo injection (Placebo Comparator)
  Interventions: Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: botulinum toxin type A — Botulinum toxin type A 75U dissolved in 3mL physiological serum injection in the upper esophageal sphincter
  Arms: Botulinum toxin injection
Drug: Sodium Chloride 0.9% Inj — Placebo: physiological serum 3mL injection in the upper esophageal sphincter
  Arms: Placebo injection

SUMMARY:
The aim of this study is to assess the effect of botulinum toxin injection into the upper esophageal sphincter in a double blind, placebo controlled study. Investigators want to assess the effect on symptoms short term (1-20 weeks after BT injection), and long term (48 weeks after BT injection).

This is a prospective double-blind randomized placebo-controlled study. Questionnaires assessing symptoms will be filled out on several occasions. At 20 weeks, a reassessment of symptoms will be done, without unblinding patients or investigator. Failures (to BT or placebo, defined as no clinical improvement or improvement less than 50%) will get the chance to receive a second procedure with active treatment (BT) in open label.

ELIGIBILITY:
Participants eligible for inclusion in this Trial must meet all of the following criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
3. Between 18 and 65 years old
4. Inability to belch, which is bothersome enough to consider treatment*, present for at least 6 months prior to inclusion, and in fulfillment of both categories a and b below:,

   1. presence of associated gastrointestinal symptoms such as abdominal bloating and discomfort/nausea, flatulence, gurgling noises from the chest or lower neck.
   2. Absence of other pharyngeal and esophageal pathologies, determined on the basis of history taking and diagnostic tests.
5. Typical findings on high resolution impedance manometry with belch provocation test (10). These typical findings include: No relaxation upon gastroesophageal gas reflux, no air clearance via the UES but instead an increased air presence time include air entrapment and oscillations.

   * Bothersome = severe enough to impact on usual activities, according to the Rome IV diagnostic criteria (11, 12).

Participants eligible for this Trial must not meet any of the following criteria:

1. Participant has a history of surgery in the upper GI tract, that might interfere with the belch reflex (such as anti-reflux surgery)
2. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
3. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial, to be decided at the discretion of the investigator.
4. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential (WOCBP) and not using an adequate, highly effective contraceptive
5. Participation in another interventional Trial with an investigational medicinal product (IMP) or device
6. >65 years old; < 18 years of age
7. Known hypersensitivity to botulinum toxin type A or to human albumin or sodium chloride
8. Presence of infection at the proposed injection site(s).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Response to Botox versus placebo, 12 weeks after treatment. | week 12
  This questionnaire is a treatment effect measure specific for inability to belch, where the change in symptoms from baseline is assessed, on a scale from 0% to 100%. 100% means complete resolution of symptoms, 0% means no improvement.

SECONDARY OUTCOMES:
Response to botox versus placebo 48 weeks after treatment. | 48 weeks
  We will use the questionnaire of 'Difficulties with belching', and response is defined as at least a 50% improvement on question 6A 'To what extent have the symptoms of 'difficulty burping air' been reduced after treatment?'.
Safety: count of each type of (serious) adverse events in each group | 4 weeks
  Safety: assessed by the number and type of (serious) adverse events that occurred in each group by week 48
Safety on swallowing: with SSQ | 4 weeks
  assessed by the Sydney Swallow Questionnaire 1 week and 4 weeks after the procedure.

OTHER OUTCOMES:
HRQOL | 1 to 48 weeks
  HRQOL using EQ-5D VAS score short-term (1, 4,12 weeks) and long-term (20 - 48 weeks after the procedure).
Patients experience and satisfaction of the treatment using overall treatment effect | 1-48 weeks
  Patients experience and satisfaction of the treatment based on OTE short-term (1, 4, 12 weeks after the procedure), and long-term (20 - 48 weeks after the procedure) OTE is an outcome measure with 9 choices: going from -4: it has become insupportable, in the middle 0: unchanged, and at the end +4: the symptoms have completely resolved.
Patients experience and satisfaction of the treatment using overall symptom severity | 1-48 weeks
  Patients experience and satisfaction of the treatment based on OSS short-term (1, 4, 12 weeks after the procedure), and long-term (20 - 48 weeks after the procedure)
Evolution of associated abdominal bloating using a VAS score for symptom severity | 1-48 weeks
  Evolution of associated abdominal bloating short-term (1, 4, 12 weeks) and long-term (20 - 48 weeks after the procedure).
Evolution of associated abdominal/thoracic pain using a VAS score for symptom severity | 1-48 weeks
  Evolution of associated abdominal/thoracic pain short-term (1, 4, 12 weeks) and long-term (20 - 48 weeks after the procedure).
Evolution of associated flatulence using a VAS score for symptom severity | 1-48 weeks
  Evolution of associated flatulence short-term (1, 4, 12 weeks) and long-term (20 - 48 weeks after the procedure).
Evolution of associated gurgling noises using a VAS score for symptom severity | 1-48 weeks
  Evolution of associated gurgling noises short-term (1, 4, 12 weeks) and long-term (20 - 48 weeks after the procedure).
Safety during follow-up, with SSQ at week 12, 20 and 48. | 12-48 weeks
  Safety during follow-up, with SSQ at week 12, 20 and 48.
Change in objective measurement of UES pressure upon belching during high resolution impedance manometry | 20 weeks
  Change in objective measurements after, versus before BT injeciton using high resolution impedance manometry at week 20, and comparing with baseline.
Change in objective measurement of oscillatory movement of air during high resolution impedance manometry | 20 weeks
  Change in objective measurements after, versus before BT injeciton using high resolution impedance manometry at week 20, and comparing with baseline.
Improvement of symptoms not reaching primary outcome | 48 weeks
  Improvement in symptoms after Botox versus placebo, 12 and 48 weeks after treatment. We will use the questionnaire of 'Difficulties with belching', using a cut-off for improvement of 30% on question 6A 'To what extent have the symptoms of 'difficulty burping air' been reduced after treatment?'.

CONTACTS AND LOCATIONS:
Overall Officials: Kathelijne G Delsupehe, MD, Principal Investigator — AZ Delta
Locations (1):
- AZ Delta, Roeselare, Belgium